CLINICAL TRIAL: NCT02247297
Title: Analysis of Serum Pancreatic Stone Protein (PSP) in Healthy Pregnant Women and Its Value in Predicting Inflammatory Complications During Pregnancy
Brief Title: Pancreatic Stone Protein (PSP) in Pregnant Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nicole Ochsenbein (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Nicole Ochsenbein, Prof. Dr. med., University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: KEK-ZH-Nr. 2014-0046
Record Dates: First submitted 2014-09-17; First posted 2014-09-25 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Pregnancy; HELLP Syndrome; Preterm Premature Rupture of Fetal Membranes; Preeclampsia
Keywords: Pancreatic stone protein (PSP); premature rupture of membranes (PPROM); amniotic infection syndrome (AIS); hemolysis, elevated liver enzymes, and low platelets (HELLP); preeclampsia; pregnancy
MeSH Terms: conditions — HELLP Syndrome; Fetal Membranes, Premature Rupture; Pre-Eclampsia; Hemolysis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant Women: Healthy pregnant women and women with preeclampsia, HELLP syndrom, amniotic infection syndrome, or preterm premature rupture of membranes
  Interventions: Procedure: Blood collection

INTERVENTIONS:
Procedure: Blood collection — Diagnostic blood collection

SUMMARY:
This prospective, single centred cohort study evaluates the physiological course of the potentially novel biomarker PSP in pregnant women as well as its predictive role in the development of inflammatory complications during pregnancy.

DETAILED DESCRIPTION:
Pregnant women feature a complex immunological condition caused by pregnancy itself and hence women present with an increased susceptibility to some infectious and non-infectious inflammatory diseases. Specifically regulated mechanisms have been described occurring in normal whereas lacking in pathological pregnancies in both the native and adaptive immune system in animal models and humans. However, clinically relevant biomarker associated with preterm premature rupture of membranes (PPROM), amniotic infection syndrome (AIS) as well as pregnancy associated complications such as preeclampsia and hemolysis, elevated liver enzymes, and low platelets (HELLP) syndrome have their limitations.

Pancreatic stone protein (PSP), originally obtained from human pancreatic stones from patients operated for chronic calcifying pancreatitis, has been studied in several gastrointestinal pathologies.

The aim of this study is to evaluate the physiological course of the potentially novel biomarker PSP in pregnant women as well as to assess its predictive role in the development of inflammatory complications during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Healthy women with single pregnancy
* Women with PPROM, AIS, preeclampsia, or HELLP syndrome
* Patients able to provide informed consent

Exclusion Criteria:

* Viral (hepatitis B virus, hepatitis C virus, human immunodeficiency virus) or confirmed bacterial infections

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women (healthy or with preeclampsia, HELLP syndrome, amniotic infection syndrome, or PPROM)
Sampling Method: Non-Probability Sample
Enrollment: 486 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Physiological course of PSP in healthy pregnant women | 34 weeks
  Measurement of serum PSP through ELISA (Enzyme Linked Immunosorbent Assay)

SECONDARY OUTCOMES:
Predictive role of PSP in the development of complications during pregnancy | 34 weeks
  Measurement of serum PSP through ELISA (Enzyme Linked Immunosorbent Assay)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Ochsenbein, Prof. Dr., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Result] De Caro A, Lohse J, Sarles H. Characterization of a protein isolated from pancreatic calculi of men suffering from chronic calcifying pancreatitis. Biochem Biophys Res Commun. 1979 Apr 27;87(4):1176-82. doi: 10.1016/s0006-291x(79)80031-5. No abstract available. PMID 111670
- [Result] Graf R, Schiesser M, Reding T, Appenzeller P, Sun LK, Fortunato F, Perren A, Bimmler D. Exocrine meets endocrine: pancreatic stone protein and regenerating protein--two sides of the same coin. J Surg Res. 2006 Jun 15;133(2):113-20. doi: 10.1016/j.jss.2005.09.030. Epub 2005 Dec 19. PMID 16360171
- [Result] Keel M, Harter L, Reding T, Sun LK, Hersberger M, Seifert B, Bimmler D, Graf R. Pancreatic stone protein is highly increased during posttraumatic sepsis and activates neutrophil granulocytes. Crit Care Med. 2009 May;37(5):1642-8. doi: 10.1097/CCM.0b013e31819da7d6. PMID 19325491
- [Result] Boeck L, Graf R, Eggimann P, Pargger H, Raptis DA, Smyrnios N, Thakkar N, Siegemund M, Rakic J, Tamm M, Stolz D. Pancreatic stone protein: a marker of organ failure and outcome in ventilator-associated pneumonia. Chest. 2011 Oct;140(4):925-932. doi: 10.1378/chest.11-0018. Epub 2011 Aug 11. PMID 21835904
- [Result] Que YA, Delodder F, Guessous I, Graf R, Bain M, Calandra T, Liaudet L, Eggimann P. Pancreatic stone protein as an early biomarker predicting mortality in a prospective cohort of patients with sepsis requiring ICU management. Crit Care. 2012 Jul 2;16(4):R114. doi: 10.1186/cc11406. PMID 22748193